CLINICAL TRIAL: NCT02999685
Title: Home-based Health Management of COPD Patients
Brief Title: Home-based Health Management of Chronic Obstructive Lung Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Minnesota HealthSolutions (Industry)
Responsible Party: Principal Investigator, Roberto P. Benzo, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-009016
Record Dates: First submitted 2016-09-29; First posted 2016-12-21 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema; Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home-base Pulm Rehab w/ Health Coaching (Active Comparator): The intervention group starts with 8 weeks of Home-base Pulmonary Rehab with Health Coaching, followed by 8 weeks of observation.
  Interventions: Behavioral: Home-base Pulmonary Rehab with Health Coaching
- Control/Wait (Active Comparator): The Control/Wait group starts with 8 weeks of observation, followed by 8 weeks of intervention (Home-base Pulm Rehab w/ Health Coaching).
  Interventions: Behavioral: Home-base Pulmonary Rehab with Health Coaching

INTERVENTIONS:
Behavioral: Home-base Pulmonary Rehab with Health Coaching

SUMMARY:
Regular physical activity has been found to be important in maintaining health and well-being in people with COPD. The purpose of this study is to test new technology and health coaching aimed to help people with COPD become more physically active in their daily lives.

DETAILED DESCRIPTION:
This study consists of a home-based pulmonary rehabilitation system. The system consists of a tablet computer, pulse oximeter, activity monitor and weekly telephone health coach calls. The rehabilitation period lasts 8 weeks. This is a randomized trial with two groups. Group A will complete the study activities during the first 8 weeks of the study followed by a period of observation. Group B will complete 8 weeks of observation followed by 8 weeks of rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* • Men and women age 40 years and older

  * Current or former smoker of at least 10 pack-years
  * Diagnosis of Global Initiative for Chronic Lung Disease (GOLD) stage II, III or IV COPD as documented by pulmonary function
  * Are eligible for Pulmonary Rehabilitation

Exclusion Criteria:

* • Unable to perform mild exercises

  * Patients with a high likelihood of being lost to follow-up or contact (patients with active chemical dependency), are planning to move out of the state, are not living in the healthcare area.
  * Patients with an inability to provide good data or follow commands (patients who are disoriented, have a severe neurologic or psychiatric condition).

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life: Chronic Respiratory Questionaire | 8 weeks from the start of the intervention
  To determine the effect of the proposed system on disease specific quality of life. The instrument has 2 summary scores, physical and emotional
Daily Physical Activity measured by Actigraph | 8 weeks from the start of the intervention
  To determine the effectiveness of the proposed system, on daily physical activity measured by triaxial accelerometers

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Benzo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benzo RP, Kramer KM, Hoult JP, Anderson PM, Begue IM, Seifert SJ. Development and Feasibility of a Home Pulmonary Rehabilitation Program With Health Coaching. Respir Care. 2018 Feb;63(2):131-140. doi: 10.4187/respcare.05690. Epub 2017 Oct 24. PMID 29066590
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials